CLINICAL TRIAL: NCT02505035
Title: Default Palliative Care Consultation for Seriously Ill Hospitalized Patients
Brief Title: Randomized Evaluation of Default Access to Palliative Services
Acronym: REDAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 822134; UH2AG050311 (NIH)
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: COPD; ESRD; Dementia
Keywords: Palliative care; Pragmatic trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Kidney Failure, Chronic; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Default ordering of palliative consult (Active Comparator): Hospitals randomized to the intervention arm will adopt a system whereby eligible patients are identified by the electronic health record, a consultation is ordered by default, and physicians may cancel the order after being alerted to it, and patients or family members may decline such services.
  Interventions: Behavioral: Default ordering of palliative consult
- Usual care (No Intervention): There will be no trial-driven approach to care. Inpatient palliative care consultative services will be actively requested by physicians as in usual care.

INTERVENTIONS:
Behavioral: Default ordering of palliative consult
  Arms: Default ordering of palliative consult

SUMMARY:
This is a large pragmatic, randomized controlled trial to test the real-world effectiveness of inpatient palliative care consultative services in improving a number of patient- and family-centered processes and outcomes of care among seriously ill hospitalized patients. The investigators hypothesize that improved patient-centered outcomes can be achieved without higher costs by simply changing the default option for inpatient palliative care consultation for eligible patients from an opt-in to an opt-out system. To test this hypothesis the investigators will conduct a clinical trial at 11 hospitals using the same electronic health record within Ascension Health, the largest non-profit health system in the U.S.

DETAILED DESCRIPTION:
The REDAPS trial aims to generate large-scale, experimental evidence regarding the real-world effectiveness of inpatient palliative consultative services (IPCS) and to test the incremental effectiveness and costs of a simple, scalable method to increase IPCS utilization among properly selected patients. The REDAPS trial will also compare the effectiveness of different palliative care team structures and services and identify patient subgroups most likely to benefit from IPCS. To achieve these goals, the investigators will conduct a clinical trial at 11 Ascension Health hospitals using the same electronic health record. Participating hospitals first contribute a minimum of 4 months of data under the control paradigm (opt-in model), where physicians must identify patients who may benefit from palliative care consultation and actively order such services. Then, using a stepped-wedge design, the hospitals are randomly assigned to begin the intervention in intervals spaced approximately 2.7 months apart. During the intervention, patients meeting consensus criteria for eligibility for palliative care consultation are identified by the electronic health record, a consultation is ordered by default, physicians may cancel the order after being alerted to it, and patients or family members may decline such services. By the end of the trial, all hospitals will have utilized the intervention paradigm of palliative care consultation for at least 4 months. The REDAPS trial will compare outcomes (clinical, economic, and process measures) before and after implementation within hospitals, as well as comparisons among hospitals at given time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. Current hospitalization of at least 3 calendar days (modified ITT)
3. Diagnosis of one or more of the following:

   * End-stage renal disease (ESRD) on dialysis
   * Chronic obstructive pulmonary disease (COPD) with home oxygen dependence or 2 or more hospitalizations in the past 12 months
   * Dementia admitted from a long-term care facility or prior placement of a surgical feeding tube or 2 or more additional hospitalizations in the past 12 months

Exclusion criteria:

1. Patients younger than 65 years old will not receive the intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34239 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Composite Measure: Length of Stay and In-Hospital Mortality | Duration of hospital stay, an expected average of 8 days
  The primary outcome is a composite measure of in-hospital mortality and hospital length-of-stay that ranks deaths along the length-of-stay distribution. Data is extracted from the electronic health record.

SECONDARY OUTCOMES:
Goals of care assessment | Duration of hospital stay, an expected average of 8 days
  Documented assessments of patients' goals of care within the electronic health record
Pain assessment | Duration of hospital stay, an expected average of 8 days
  Documented assessments of patients' pain scores within the electronic health record
Dyspnea assessment | Duration of hospital stay, an expected average of 8 days
  Documented assessments of patients' dyspnea within the electronic health record
Code status | Duration of hospital stay, an expected average of 8 days
  Code status documented within the electronic health record
Mechanical ventilation | Duration of hospital stay, an expected average of 8 days
  Documented orders for mechanical ventilation within the electronic health record
Cardiopulmonary resuscitation | Duration of hospital stay, an expected average of 8 days
  Documented orders for cardiopulmonary resuscitation within the electronic health record
Inpatient dialysis | Duration of hospital stay, an expected average of 8 days
  Documented orders for dialysis during inpatient stay within the electronic health record
ICU admission | Duration of hospital stay, an expected average of 8 days
  Transferal to an intensive care unit documented within the electronic health record
Hospital discharge status | Duration of hospital stay, an expected average of 8 days
  Hospital discharge disposition code documented within the electronic health record
Discharge planning orders | Duration of hospital stay, an expected average of 8 days
  Discharge orders for home care services documented within the electronic health record
Hospital readmission | 30 days
  30-day hospital re-admissions documented within the Premier database
Direct cost per day | Duration of hospital stay, an expected average of 8 days
  Direct cost per day documented within the Premier database
Direct cost per hospitalization | Duration of hospital stay, an expected average of 8 days
  Direct cost per hospitalization documented within the Premier database

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, PhD,MD, Principal Investigator — University of Pennsylvania
Locations (11):
- United States (11):
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - St. Vincent's Medical Center, Riverside, Jacksonville, Florida
  - St. Vincent's Medical Center, Southside, Jacksonville, Florida
  - Via Christi Hospital, St. Francis, Wichita, Kansas
  - Via Christi Hospital, St. Joseph, Wichita, Kansas
  - Borgess Medical Center, Kalamazoo, Michigan
  - Our Lady of Lourdes Memorial Hospital, Binghamton, New York
  - St. Thomas West Hospital, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Columbia St. Mary's, Ozaukee, Mequon, Wisconsin
  - Columbia St. Mary's, North Lake, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Courtright KR, Madden V, Bayes B, Chowdhury M, Whitman C, Small DS, Harhay MO, Parra S, Cooney-Zingman E, Ersek M, Escobar GJ, Hill SH, Halpern SD. Default Palliative Care Consultation for Seriously Ill Hospitalized Patients: A Pragmatic Cluster Randomized Trial. JAMA. 2024 Jan 16;331(3):224-232. doi: 10.1001/jama.2023.25092. PMID 38227032
- [Derived] Courtright KR, Madden V, Gabler NB, Cooney E, Small DS, Troxel A, Casarett D, Ersek M, Cassel JB, Nicholas LH, Escobar G, Hill SH, O'Brien D, Vogel M, Halpern SD. Rationale and Design of the Randomized Evaluation of Default Access to Palliative Services (REDAPS) Trial. Ann Am Thorac Soc. 2016 Sep;13(9):1629-39. doi: 10.1513/AnnalsATS.201604-308OT. PMID 27348271